CLINICAL TRIAL: NCT05507151
Title: Effectiveness of Endoscopic Sleeve Gastroplasty in Obese Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Effectiveness of Endoscopic Sleeve Gastroplasty in Nonalcoholic Fatty Liver Disease/Nonalcoholic Steatohepatitis
Status: Recruiting | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Shailendra Singh, Associate Professor, West Virginia University
Other Study IDs: 2202523300
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic Sleeve Gastroplasty: endoscopic suturing of the stomach
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty

INTERVENTIONS:
Procedure: Endoscopic Sleeve Gastroplasty — endoscopic suturing of the stomach

SUMMARY:
Endoscopic weight loss procedures, also termed endoscopic sleeve gastroplasty (ESG), has been proposed as a non-surgical procedure for managing obesity and offers a standard weight loss approach. Realizing there is a knowledge gap in applying ESG to morbidly obese patients with NAFLD, the investigators propose studying the efficacy of weight control and functional outcomes of ESG. This prospective pilot study is aimed to study the safety profiles, quality of life, and changes and improvements in the anthropometric, metabolic, and biochemical changes in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m2, who are eligible for ESG
* Patients scheduled to undergo an endoscopic bariatric weight loss procedure (ESG)
* Patients older than 18 years and younger than 75 years of age at the time of consent
* Patients able to provide written informed consent on the Institutional review board (IRB) approved informed consent form
* Patients willing and able to comply with study requirements for follow-up

Exclusion criteria:

* Patients who are treated with intragastric balloons
* Family history of esophageal, gastric, or duodenal malignancy and active gastric ulceration,
* Pre-existing esophageal stenosis/stricture preventing the advancement of an endoscope during screening/baseline Esophagogastroduodenoscopy (EGD)
* Presence of any gastric condition which required endoscopic surveillance (e.g., known gastric intestinal metaplasia),
* Known vascular abnormalities, obligate therapeutic anticoagulation, and pregnancy/lactation
* Evidence of end-stage liver disease, including portal hypertension, ascites, and coagulopathy
* Positivity for hepatitis B virus or hepatitis C virus, current alcohol consumption of more than 20 g/day in females and more than 30 g/day in males on average, use of medications with reported hepato-steatogenic effect (amiodarone, tamoxifen, estrogens), and drug-induced liver disease
* Type 1 diabetes, Prior bariatric surgery, Autoimmune liver disease (antinuclear antibody titer >1/160), Wilson's disease, hemochromatosis, alpha1-antitrypsin deficiency,
* Known positivity for human immunodeficiency virus, a concomitant disease with reduced life expectancy, severe psychiatric condition, drug dependence, or inability to provide informed consent.
* The patient refuses or is unable to provide written informed consent
* Prior bariatric treatment procedure

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 obese patients undergoing an endoscopic sleeve gastroplasty (ESG).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Controlled Attenuation Parameter of Steatosis | Baseline (Before ESG)
  The CAP measures ultrasonic attenuation in the liver at 3.5 MHz using signals acquired by the FibroScan® M probe based on vibration-controlled transient elastography. The final CAP value, which ranges from 100 to 400 decibels per metre (dB/m), is the median of individual measurements. Higher measure indicates higher portion of liver affected by fatty change.
Change in Controlled Attenuation Parameter of Steatosis | 6 months post ESG
  The CAP measures ultrasonic attenuation in the liver at 3.5 MHz using signals acquired by the FibroScan® M probe based on vibration-controlled transient elastography. The final CAP value, which ranges from 100 to 400 decibels per metre (dB/m), is the median of individual measurements. Higher measure indicates higher portion of liver affected by fatty change.
Change in Controlled Attenuation Parameter of Steatosis | 12 months post ESG
  The CAP measures ultrasonic attenuation in the liver at 3.5 MHz using signals acquired by the FibroScan® M probe based on vibration-controlled transient elastography. The final CAP value, which ranges from 100 to 400 decibels per metre (dB/m), is the median of individual measurements. Higher measure indicates higher portion of liver affected by fatty change.
Change in Liver Stiffness Measurement of Fibrosis | Baseline (Before ESG)
  Liver stiffness result is measured in kilopascals (kPa) Range is 0-75kPa. Normal results are usually between 2 and 7 kPa. The highest possible result is 75 kPa. Higher results indicate liver disease.
Change in Liver Stiffness Measurement of Fibrosis | 6 months post ESG
  Liver stiffness result is measured in kilopascals (kPa) Range is 0-75kPa. Normal results are usually between 2 and 7 kPa. The highest possible result is 75 kPa. Higher results indicate liver disease.
Change in Liver Stiffness Measurement of Fibrosis | 12 months post ESG
  Liver stiffness result is measured in kilopascals (kPa) Range is 0-75kPa. Normal results are usually between 2 and 7 kPa. The highest possible result is 75 kPa. Higher results indicate liver disease.

SECONDARY OUTCOMES:
Anthropometric Evaluation | 6 months post ESG
  Changes in Anthropometric evaluation from baseline to 6 months post ESG
BMI Changes | 6 months post ESG
  Compare the change in BMI from baseline to the 6 months post ESG. Body Mass Index (BMI) is a person's weight in kilograms (or pounds) divided by the square of height in meters (or feet).
BMI Changes | 12 months post ESG
  Compare the change in BMI from baseline to the 12 months post ESG. Body Mass Index (BMI) is a person's weight in kilograms (or pounds) divided by the square of height in meters (or feet).
Excess Weight Loss Changes | 6 months post ESG
  Percent excess weight loss change from baseline to 6 months
Excess Weight Loss Changes | 12 months post ESG
  Percentage of excess weight loss change from baseline to 12 months
Total Body Weight Loss Changes | 6 months post ESG
  Percentage of total body weight loss (TBWL) from baseline to 6 months
Total Body Weight Loss Changes | 12 months post ESG
  Percentage of total body weight loss (TBWL) from baseline to 12 months
Absolute Body Weight Loss Changes | 6 months post ESG
  Percentage of Absolute Body Weight Loss from baseline to 6 months
Absolute Body Weight Loss Changes | 12 months post ESG
  Percentage of Absolute Body Weight Loss from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shailendra Singh, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States